CLINICAL TRIAL: NCT05061433
Title: Mobile Integrated Healthcare and Community Paramedicine: A Pilot Project Using LifePACT Critical Care Physician, Paramedic, and RN Staff to Increase Patient Satisfaction and Reduce Hospital Readmissions
Brief Title: Mobile Integrated Healthcare and Community Paramedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 693277
Record Dates: First submitted 2021-09-21; First posted 2021-09-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-09

CONDITIONS: Hospital Readmission; Pneumonia; Myocardial Infarction; COPD
MeSH Terms: conditions — Pneumonia; Myocardial Infarction; Pulmonary Disease, Chronic Obstructive | interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants receive standard of care.
- Intervention (Experimental): Initial Home Visit: MIH/CP provider team will visit the patient's home at the scheduled time following a specific General Followup Protocol involving 1. Assessment of patient understanding of recent illness and medical therapy including reinforcement of medical adherence, 2. Any other disease-specific concerns, 3. Performance of a home safety evaluation, 4. If patients have concerns relating to their ability to manage their disease process at home, 5. MIH/CP providers and an on-call social worker will provide assistance in the form of on-site, telephone, and electronic referrals or provision of appointments with appropriate services.
  Subsequent visits: The MIH/CP team will decide in conjunction with Medical Control and the PMD if further followup is needed, and the most appropriate followup interval., At 30 days from initial hospital discharge, the patient will be discharged from the MIH/CP program in conjunction with the PMD.
  Interventions: Other: Mobile Integrated Healthcare/Community Paramedicine (MIH/CP) Support

INTERVENTIONS:
Other: Mobile Integrated Healthcare/Community Paramedicine (MIH/CP) Support — MIH/CP provider and their team will offer additional support and connection to resources after patient is discharged from hospital.
  Arms: Intervention

SUMMARY:
Background:

Initially conceived of as a method to address healthcare needs of underserved rural populations, Mobile Integrated Healthcare and Community Paramedicine (MIH/CP) is a new model of inter-professional, community-based outpatient healthcare delivery that primarily utilizes the resources and training of Emergency Medical Services (EMS) to fill gaps in local healthcare infrastructure, expanding existing scope of practice in most cases while not detracting from acute transport capabilities.

Although programs have been in existence since the early 1990s, there are few objective studies of the efficacy, safety, and cost-effectiveness of MIH/CP programs, many of which are limited-scope pilot projects. The limited data already published on these measures by established programs shows substantial Medicare charge-avoidances in patients enrolled in CHF-readmission prevention and EMS frequent user programs, and a significant reduction in Emergency Department visits overall, especially in austere environments.

In summary, MIH/CP is an attempt at formalization of long-standing practices to collaborate with and supplement other healthcare system components such as primary care and home health services. Standardized, objective data collection and publication of results will be needed to support continuation and financial support of this emerging concept.

Objective/Hypothesis:

Using the existing resources of the MD-, RN- and Paramedic-staffed Lifespan Pediatric and Adult Critical Care Transport (LifePACT) service, investigators aim to study whether implementation of an MIH/CP pilot program tailored to the needs of an urban, underserved population in Providence, Rhode Island, will reduce the rate of 30-day hospital readmissions for patients after discharges for community-acquired pneumonia, acute MI, and COPD. In addition, investigators will study whether such a program is considered to be safe (in terms of not increasing the number of adverse events post-discharge for patients or compromising the efficacy of the LifePACT transport role) and considered satisfactory by patients (rated comparably to visits by other outpatient health care services such as VNA services).

ELIGIBILITY:
Inclusion Criteria:

* Current inpatient/observation status for: NSTEMI; CHF; PNA (community or HCAP); COPD; Wound infection or complication,
* English Speaking,
* Not pregnant,
* Not incarcerated,
* Able to maintain clinical sobriety for informed consent and home visitation.,
* No unstable psychiatric conditions (Patients may be under treatment for mental health conditions as long as their symptoms are controlled).,
* Accessible and reliable place of residence that is not a nursing home or "on the street" location. (Homeless patients are eligible as long as they have consistent access to a domicile that can provide shelter and privacy).,
* No anticipated VNA or home care within 24-36 hours of visit,
* Ages 18-80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital readmissions | 30 days
Incidence of adverse medical events | 30 days
Incidence of ED visits | 30 days

IPD SHARING:
Plan to Share IPD: Undecided